CLINICAL TRIAL: NCT03351309
Title: Telephone Cognitive Behavioral Therapy for Veterans Undergoing Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Iowa City Veterans Affairs Medical Center (U.S. Federal Agency)
Collaborators: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Principal Investigator, Katherine Hadlandsmyth, Clinical Assistant Professor of Anesthesia - Chronic Pain Medicine, Iowa City Veterans Affairs Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 201708823
Record Dates: First submitted 2017-11-02; First posted 2017-11-22 (Actual); Last update posted 2021-08-24 (Actual); Status verified 2021-08

CONDITIONS: Persistent Post-surgical Pain; Veterans

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Telephone-based cognitive behavioral therapy (Experimental): Telephone-based cognitive behavioral therapy (CBT) intervention - Four session protocol plus routine perioperative management.
  Interventions: Behavioral: Telephone-based Cognitive Behavioral Therapy (CBT)
- Treatment as Usual (No Intervention): Treatment as Usual (TAU) - Routine perioperative management.

INTERVENTIONS:
Behavioral: Telephone-based Cognitive Behavioral Therapy (CBT) — Four session telephone CBT protocol.
  Arms: Telephone-based cognitive behavioral therapy

SUMMARY:
The study team propose to investigate the feasibility and pilot a Telephone Cognitive Behavioral Therapy intervention for those identified to be at risk for chronic pain following surgery.

ELIGIBILITY:
Inclusion Criteria:

1) >18 years of age, 2) scheduled for hernia repair, breast surgery, amputation, thoracotomy, cholecystectomy, cardiac surgery, splenectomy, orthopedic, urological or vascular surgery, 3) Rural dwelling

Exclusion Criteria:

1) language or cognitive barriers preventing completion of questionnaires, 2) severe psychiatric disorder: bipolar or psychotic disorder, 3) significant surgical complications.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2017-11-25 (Actual); Primary Completion 2021-08-01 (Actual); Study Completion 2021-08-01 (Actual)

PRIMARY OUTCOMES:
Pain Severity | 3 months post-surgery
  Numeric Rating Scale of surgical site pain: none-mild (0-3) compared to Moderate-severe (4+)

SECONDARY OUTCOMES:
Qualitative analysis of feasibility data | Between 1-2 weeks post-TCBT
  Qualitative interviews with a subset of TCBT participants, until data saturation is reached.
Pain severity - continuous | 3 months post-surgery
  Brief Pain Inventory
Pain-related functioning | 3 months post-surgery
  Pain Disability Index
Opioid and other analgesic use | 3 months post-surgery
  Self-report medication use
Depression | 3 months post-surgery
  Patient Health Questionnaire
Anxiety | 3 months post-surgery
  Generalized Anxiety Disorder Scale
  * Generalized Anxiety Disorder 7-item (GAD-7) scale measures endorsement/symptoms of generalized anxiety.
  * The scores for each individual question range from 0 to 3 (0 = not at all, 1 = several days, 2 = more than half the days, 3 = nearly every day). A total score can range from 0-21.
  * A score of 5 is a cut-off for mild anxiety, 10 is a cut-off for moderate anxiety, and 15 is a cut-off for severe anxiety. Higher values represent worse outcomes.
  * To compute a total score, all items with endorsements of 1 or greater are added together for a composite score of 0-21.
Health-related quality of life: SF-36 | 3 months post-surgery
  SF-36
  * 36-Item Short Form Survey Instrument (SF-36) measures eight constructs related to quality of life:
    * Physical functioning
    * Role limitations due to physical health
    * Role limitations due to emotional problems
    * Energy/fatigue
    * Emotional well-being
    * Social functioning
    * Pain
    * General health
  * Each item is recoded to reflect score ranges from 0 to 100 where 0 is the least favorable and 100 is the most favorable. Each item corresponds to a specific construct. Items associated with each construct are averaged to retrieve a construct score. Scores are then converted into z-scores.
  * Higher z-scores reflect a more favorable health status.
Patient satisfaction with outcomes | 3 months post-surgery
  Brief satisfaction items regarding TCBT intervention (Only for participants assigned to receive TCBT)
  1. Overall, how satisfied are you with the TCBT? (very dissatisfied, dissatisfied, neutral, satisfied, very satisfied)
  2. How satisfied are you with the TCBT for reducing your pain or helping you cope with your pain? (very dissatisfied, dissatisfied, neutral, satisfied, very satisfied)
  3. How satisfied are you with the TCBT for improving your functioning? (very dissatisfied, dissatisfied, neutral, satisfied, very satisfied).

CONTACTS AND LOCATIONS:
Overall Officials: Katherine Hadlandsmyth, Ph.D., Principal Investigator — University of Iowa
Locations (1):
- Iowa City VA Medical Center, Iowa City, Iowa, United States